CLINICAL TRIAL: NCT02162238
Title: Assessment of Zinc Intake From Enriched Water and Other Dietary Sources in Kisumu, Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: ETH Zurich (Other); Maseno University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Kisumu dietary Zn Study
Record Dates: First submitted 2014-04-16; First posted 2014-06-12 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Zinc Deficiency
Keywords: zinc; diet; water; morbidity; growth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- purified water (Placebo Comparator): Filtered water Pump water purified by the LSF-filtering device Intervention: Device: LSF-filtering device
- zinc enriched purified water (Experimental): Zinc water water purified and zinc-enriched by the LSF-filtering device Intervention: Device: LSF-filtering device
  Interventions: Device: LSF-filtering device

INTERVENTIONS:
Device: LSF-filtering device — Device: LSF-filtering device LifeStraw Family is a water purification device that by means of hollow fibres removes solid particles (<0.5 Nephelometric Turbidity units turbidity reduction), bacteria (>Log 6 reduction), viruses (>Log 4 reduction) and cysts (>Log 3 reduction). Zinc enrichment is provided by a chamber housing a zinc releasing glass-plate that is placed annexed to the hollow fibre column. It is estimated that the LSF can provide about 5 mg of zinc/l of filtered water. By consuming daily a portion of 0.6 litres of enriched water, >100% of the age-specific estimated physiologic requirement would be covered, assuming a fractional absorption of 40%.
  Other Names: LifeStraw Family by Vestergaard Frandsen SA
  Arms: zinc enriched purified water

SUMMARY:
Introduction: The prevalence of low serum zinc in children under 5 in East Seme, Kisumu is 73.5% and this is likely due at least in part to low bioavailable zinc from the local cereal-based diet. Interventions that will increase zinc intake could prove useful in the effort to control zinc deficiency. A potential strategy is to increase zinc intake through enriched or fortified water. The Life Straw Family filter (LSF, Verstergaard Frandsen S.A, Switzerland) is capable of purifying water and at the same time enriching it with zinc at a variable concentration with mean delivery of approximately 1-4mg/L.

Aims of the study: The primary aim of this study will be to quantify in under 5 year old children the contribution of the household LSF device to zinc intake and dietary zinc bioavailability in participating households. Secondary objectives are; 1) to assess change in serum zinc levels, growth, morbidity in the intervention group compared to control; 2) to characterize composition of the intestinal flora of children in the intervention group compared to control.

Study Design and Methods:

Consenting households from East Seme, Kisumu, Kenya will be randomly allocated to 2 treatment arms in an effectiveness study (90 under-five's per treatment arm). Group one will receive the LSF device with the zinc delivery system; group 2 will receive a LSF without the zinc delivery system.

Zinc intake will be assessed in a subsample of the under 5 year old children enrolled in the effectiveness trial (n=100). This will be estimated by 24 hr recalls administered on 2 non-consecutive days in the dry and wet season. Selected food samples will be collected for direct analysis of zinc and phytic acid content, to supplement data from food composition tables (FCT's). The dietary assessment data will be used to estimate the distribution of zinc intakes in this age group and the EAR cut-off method will be used to estimate the proportion at risk of inadequate intakes.

Data on water intake from the LSF device will be obtained by personal diaries and tally counters. The Zn concentration of the filtered water will be measured weekly. Using these data and the data from the dietary assessment, the contribution of the LSF zinc delivery to the overall dietary zinc intake will be estimated.

The effectiveness study will be conducted as a 6-month double blind randomised trial with 3 assessment time points (baseline, midpoint and endpoint). Three ml (3ml) whole blood will be collected from under 5 year old children enrolled in the households for determination of serum zinc (SZn), C-reactive protein (CRP), Alpha-1- acid glycoprotein (AGP) and hemoglobin (Hb). Stool samples will be collected from a subsample at baseline, midpoint and endpoint in the intervention and control group to assess the composition of the gut microflora and gut inflammation. Anthropometrics (weight and height) will be measured at baseline, midpoint and endpoint of the study. Weekly active surveillance for incidence and severity of malaria, diarrhea and other infectious diseases will be done by questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Children (under 5 year olds) in consenting households will participate in the study

Exclusion Criteria:

* Subjects with severe anemia (Hb<7g/dl)
* Subjects receiving zinc supplementation
* Subject with chronic diseases affecting zinc metabolism, such as kidney diseases or chronic gastrointestinal disease.
* Subjects participating in any other clinical trials in the study site

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
number of participants with adequate zinc intake above the EAR (estimated average requirement) | 6 months

SECONDARY OUTCOMES:
number of participants with increased serum zinc level from baseline | at 3 months into intervention and at 6 months
morbidity incidence | every week up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diego Moretti, PhD, Principal Investigator — ETH Zurich; Inge D Brouwer, PhD, Study Director — Wageningen University; Michael B Zimmerman, PhD, Study Chair — ETH Zurich and Wageningen University; Pauline Andango, PhD, Study Director — Maseno University
Locations (1):
- Maseno University, Kisumu, Nyanza, Kenya

REFERENCES:
- [Derived] Kujinga P, Galetti V, Onyango E, Jakab V, Buerkli S, Andang'o P, Brouwer ID, Zimmermann MB, Moretti D. Effectiveness of zinc-fortified water on zinc intake, status and morbidity in Kenyan pre-school children: a randomised controlled trial. Public Health Nutr. 2018 Oct;21(15):2855-2865. doi: 10.1017/S1368980018001441. Epub 2018 Jun 7. PMID 29877169